CLINICAL TRIAL: NCT07253155
Title: Probiotics Use and Preventing Gastrointestinal Symptoms in People Living With Overweight and Obesity.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Ferryx Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: REC/25/0042
Record Dates: First submitted 2025-09-23; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Gut Inflammation; Overweight and Obese Volunteers
Keywords: Obesity; gut inflammation; gastrointestinal symptoms; microbiota; metabolome; overweight
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blinded to participants and researchers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Arm (Experimental): Probiotic supplement arm, 2 capsules consumed/day for a period of 28 days.
  Interventions: Dietary Supplement: Probiotic Arm
- Placebo Arm (Placebo Comparator): Placebo supplement arm, 2 capsules consumed/day for a period of 28 days.
  Interventions: Dietary Supplement: Placebo Arm

INTERVENTIONS:
Dietary Supplement: Probiotic Arm — 1 x10^9 cfu Streptococcus thermophilus (FX856), corn starch, anti-caking agent in a hydroxypropylmethycellulose & pectin capsule.
  Arms: Probiotic Arm
Dietary Supplement: Placebo Arm — corn starch, anti-caking agent in a hydroxypropylmethycellulose & pectin capsule.
  Arms: Placebo Arm

SUMMARY:
Inflammatory bowel disease (IBD) affects over 6.8 million people worldwide, with current treatments often causing side effects and poor patient compliance. Dysbiosis of gut microbiota is a key factor, and while probiotics are considered safe and beneficial, conventional strains fail to function effectively during active inflammation due to high iron levels in the gut. Streptococcus thermophilus (FX856), unlike traditional probiotics, can thrive in this iron-rich environment, promoting mucosal healing. A 2-way crossover intervention study will be conducted with FX856 supplementation in overweight and obese individuals who often exhibit mild gut inflammation by measuring faecal calprotectin and systemic inflammatory markers.

DETAILED DESCRIPTION:
There is a lack of satisfactory treatments for inflammatory bowel disease (IBD), an excruciatingly debilitating condition which affects 1 in 123 people in the UK (>0.5million). Current treatments have significant negative side effects, affecting quality of life of patients and reducing compliance, leading to exacerbation of symptoms. Dysbiosis in the composition of gut microbiota is one of the leading causes of chronic inflammatory diseases such as inflammatory bowel disease (IBD). Supplementation with dietary components is a promising approach for the treatment of inflammatory bowel disease (IBD) and the use of probiotics for IBD treatment has shown promising effects on consumers' quality of life, they are popular due to their perception as safe, natural treatments but currently marketed products cannot function during active disease. Streptococcus thermophilus (FX856) is an OTC supplement already available in the UK that has a unique ability to survive and thrive during active inflammation, allowing it to promote mucosal healing in the inflamed gut, an area where conventional probiotics have failed. During active inflammation or stress, gut iron levels increase. This iron-rich environment compromises the suitability of conventional probiotic bacteria that have been, and are still, commonly trailed for the relief of symptoms in patients suffering from gut inflammation. Whilst most constituents of the gut microbiome are able to increase growth rate in response to iron, species traditionally employed as probiotics, such as lactobacilli and bifidobacteria, are unable to use iron as a growth factor; they are outcompeted under high iron conditions and cannot have a beneficial effect. Unlike most bacterial strains used as probiotics, FX856 can maintain growth within an iron-rich environment, as observed in the inflamed intestine. Faecal calprotectin is considered a suitable non-invasive surrogate marker of intestinal inflammation in inflammatory bowel disease and is reported to be increased in obese individuals. Consequently, this study will determine how the probiotic FX856 interacts with the gut and immune system to reduce inflammation. A 2-way crossover intervention study will be conducted with FX856 (4 weeks) in an overweight and obese population, as such individuals are likely to have chronic mild gut inflammation and examine markers of faecal calprotectin and circulating inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Either a BMI 25+ kg/m2 and be aged 40+ years or have a BMI 30+ kg/m2 and aged 18+ years
* Males and females (not currently pregnant/lactating)
* Omnivorous diet (consuming plant & animal based foods)
* Not taking any medication affecting the gastro-intestinal tract
* No chronic gastro-intestinal illness
* Not using fibre supplements or any probiotic or prebiotic products, e.g., Fybogel, Actimel, kefir or kimchee for at least 6 weeks prior to study
* Not consuming 7+ units of alcohol per day (e.g. 3 medium glasses of wine ~12%)

Exclusion Criteria:

* Not aged 40+ years (if have a BMI 25-29.9 kg/m2)
* BMI<30 kg/m2 (if aged 18-39 years)
* Pregnant/lactating female
* Vegan/vegetarian/high protein diet
* Chronic gastro-intestinal illness
* Taking medication affecting the gastro-intestinal tract
* Taking fibre supplements or any probiotic or prebiotic products
* Consuming 7+ units of alcohol per day (e.g. 3 medium glasses of wine ~12%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Assess effects of FX856 on faecal calprotectin | Change over 28 days comparison between treatments
  The level of calprotectin in faecal samples will be measured by immunoassay in all participants to determine if FX856 consumption can decrease it.

SECONDARY OUTCOMES:
Assess effect of FX856 treatment on gastrointestinal symptoms | Change over 28 days comparison between treatments
  Measured by questionnaire rated on scale from 0 (Dose not bother me at all) to 10 (Is as bad as I can imagine)
Assess effect of FX856 on circulating inflammatory cytokines IFN-γ | Change over 28 days comparison between treatments
  Measured by ELISA
Assess effect of FX856 on circulating inflammatory cytokines IL-1β | Change over 28 days comparison between treatments
  Measured by ELISA
Assess effect of FX856 on circulating inflammatory cytokines IL-6 | Change over 28 days comparison between treatments
  Measured by ELISA
Assess effect of FX856 on circulating inflammatory cytokines TNF-α | Change over 28 days comparison between treatments
  Measured by ELISA
Assess effect of FX856 on Cholesterol | Change over 28 days comparison between treatments
  Measured by ILab 650 chemistry analyser using CHOD-PAP/GPO-PAP colorimetric end-point assays.
Assess effect of FX856 on LDL cholesterol | Change over 28 days comparison between treatments
  Measured by ILab 650 chemistry analyser using CHOD-PAP/GPO-PAP colorimetric end-point assays. LDL concentrations calculated using the Friedewald formula.
Assess effect of FX856 on HDL cholesterol | Change over 28 days comparison between treatments
  Measured via ILab 650 chemistry analyser using CHOD-PAP/GPO-PAP colorimetric end-point assays.
Assess effects of FX856 on microbiota | Change over 28 days comparison between treatments
  The composition of gut microbiota from faecal samples will be measured by NGS pre and post consumption in all participants to determine if FX856 consumption alters the gut microbiota.
Assess effects of FX856 on faecal metabolome | Change over 28 days comparison between treatments
  The faecal metabolome from faecal samples will be measured by untargeted mass spec pre and post consumption in all participants to determine if FX856 consumption alters the faecal metabolome.
Assess effects of FX856 on blood metabolome | Change over 28 days comparison between treatments
  The blood metabolome will be measured by untargeted mass spec pre and post consumption in all participants to determine if FX856 consumption alters the blood metabolome.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Gill, PhD, Principal Investigator — Ulster University, Human Intervention Studies Unit, Coleraine, Co. Londonderry, BT52 1SA, United Kingdom.
Locations (1):
- Ulster University, Human Intervention Studies Unit, Coleraine, United Kingdom

IPD SHARING:
Plan to Share IPD: No